CLINICAL TRIAL: NCT06541158
Title: Testing the Feasibility of a Transportation for Cancer Care Navigation Tool (TRACT) in Solid Tumors Patients Receiving Radiotherapy
Brief Title: Transportation for Cancer Care Navigation Tool for Reducing Travel Barriers Among Patients With Solid Tumors Receiving Radiation Therapy
Acronym: TRACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jinbing Bai, Jinbing Bai, PhD, RN, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00007528; NCI-2024-05756 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00007528; WINSHIP6207-24 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Malignant Solid Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods; Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stage I (CAB) (Experimental): Participants meet with the study research team to develop and refine the TRACT program.
  Interventions: Other: Discussion
- Stage II Group I (TRACT program) (Experimental): Patients receive the TRACT program consisting: of 1) Screening of travel barriers; 2) Awareness of transportation obstacles and resources using videos, 3) Assistance with transportation resource application and utilization, and 4) Alignment of community resources to navigate individualized transportation support by the trained travel navigator for 3 months.
  Interventions: Behavioral: Health Promotion and Care; Other: Questionnaire Administration
- Stage II Group II (usual care, video, pamphlet) (Active Comparator): Patients receive usual care with PAF pamphlet for 3 months.
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Media Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Stage II Group II (usual care, video, pamphlet)
Other: Discussion — Participate in a CAB
  Other Names: Discuss
  Arms: Stage I (CAB)
Other: Educational Intervention — Receive PAF pamphlet
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Stage II Group II (usual care, video, pamphlet)
Behavioral: Health Promotion and Care — Receive the TRACT program
  Arms: Stage II Group I (TRACT program)
Other: Media Intervention — Receive transportation awareness brief video
  Arms: Stage II Group II (usual care, video, pamphlet)
Other: Questionnaire Administration — Ancillary studies
  Arms: Stage II Group I (TRACT program); Stage II Group II (usual care, video, pamphlet)

SUMMARY:
This clinical trial evaluates whether the Transportation for Cancer Care Navigation Tool (TRACT) can reduce travel barriers among patients with solid tumors receiving radiation therapy. It is estimated that 20-30% patients with cancer experience travel-related barriers for cancer care. This is a particular problem for patients with radiation therapy as these patients frequently receive multiple treatment cycles, which often require daily treatment for multiple weeks or months. Addressing travel barriers has been a prerequisite for cancer care as travel barriers negatively influence cancer treatment adherence and cancer care outcomes, such as survival and quality of life. The TRACT program may help reduce travel barriers and therefore promote health equity among patients with solid tumors receiving radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To work collaboratively with a Community Advisory Board (CAB, e.g., patients, caregivers, clinicians, and social workers) to refine a theory-driven TRACT program for solid tumor patients receiving radiation therapy (RT) with travel barriers.

II. To evaluate the feasibility of the TRACT program for patients with solid tumors receiving RT with travel barriers.

III. To explore the efficacy of the TRACT program on RT adherence (canceling, delaying, missing, or terminating essential care) and patient-reported outcomes (PROs) (distress, financial toxicity, and quality of life [QOL]) compared to enhanced usual care (EUC, usual care + transportation awareness brief video with Patient Advocate Foundation [PAF] pamphlet).

OUTLINE:

STAGE I (CAB): Participants meet with the study research team to develop and refine the TRACT program.

STAGE II: Patients are randomized to 2 groups.

GROUP I: Patients receive the TRACT program consisting: of 1) Screening of travel barriers; 2) Awareness of transportation obstacles and resources using videos, 3) Assistance with transportation resource application and utilization, and 4) Alignment of community resources to navigate individualized transportation support by the trained travel navigator for 3 months.

GROUP II: Patients receive usual care with PAF pamphlet for 3 months.

After completion of study intervention, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosed with solid tumors
* Undergoing RT (not excluded with chemotherapy)
* Competent to give consent
* English-speaking
* With travel barriers as screened by the reliable and validated 10-item Transportation Barriers Measure. In this study, item 2 ("how much trouble is it for you to get transportation to your doctor or treatment?") from the general barriers domain will be used to screen patients for travel barriers

Exclusion Criteria:

* Receive palliative care
* Are non-English-speaking (excluded due to pilot data without fund to support translation services)
* Are enrolled in lodging programs (e.g., the American Cancer Society [ACS] Hope Lodge®)
* Have major depression/anxiety disorders that interfere with their ability to participate (based on the electronic medical records report)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility of screening patients for the Transportation for Cancer Care Navigation Tool (TRACT) program | At T0 (pre-intervention) and T1 (3 months post-intervention)
  Will be assessed by response rates, time burden (minutes to complete the measure), and percent of positive screenings. Will use descriptive statistics. Differences between the two groups will be assessed by an independent two-sample t-test or Chi-squared test if applicable. A 95% level of statistical confidence will be assumed.
Recruitment to the TRACT program (Feasibility) | At T0 (pre-intervention) and T1 (3 months post-intervention)
  Will be assessed by the number of patients screened and randomized. Will use descriptive statistics. Differences between the two groups will be assessed by an independent two-sample t-test or Chi-squared test if applicable. A 95% level of statistical confidence will be assumed.
Retention and adherence rate (Feasibility) | At T0 (pre-intervention) and T1 (3 months post-intervention)
  Will be assessed by the total number of meetings and time spent with the travel navigator for travel resources, percentage of patients using travel resources, percentage of patients with completed measures. Differences between the two groups will be assessed by an independent two-sample t-test or Chi-squared test if applicable. A 95% level of statistical confidence will be assumed.
Acceptability of the Transportation for Cancer Care Navigation Tool | At T0 (pre-intervention) and T1 (3 months post-intervention)
  Will be assessed by the 4-item Acceptability of Intervention Measure with Cronbach alpha=0.85-0.91. Differences between the two groups will be assessed by an independent two-sample t-test or Chi-squared test if applicable. A 95% level of statistical confidence will be assumed.
Travel barriers | At T0 (3 months) and T1 (3 months post-intervention)
  Will be reported as transportation mode (e.g., public transportation, drive-myself, drive-someone else drives me), owning a car (yes/no), parking cost, and travel cost for each appointment. Travel distance and time to cancer treatment facilities will be estimated by ArcGIS 10.3. Categorical and continuous variables will be used to present this outcome variable.
Treatment adherence | At T1 (3 months post-intervention)
  Will be assessed by canceling, missing, delaying, or terminating essential care. Nonadherence rates will be calculated as the number of no-shows, same-day cancellations, delays, and early stoppage of treatment divided by the total number of treatment days based on data within the electronic health records (EMRs). A percentage of completion rate of treatment will be calculated to present the treatment adherence.
Distress | At T0 (3 months) and T1 (3 months post-intervention)
  Will be measured by the National Comprehensive Cancer Network (NCCN) Distress Thermometer. The one-item 11-point Likert scale represented on a visual graphic of a thermometer ranging from 0 (no distress) to 10 (extreme distress) will be used to assess patients' distress. Will be assessed using mixed-effect analysis of variance to model the correlations.
Financial toxicity | At T0 (3 months) and T1 (3 months post-intervention)
  Will be measured by the Comprehensive Score for Financial Toxicity (COST). The COST is a 5-point Likert scale evaluating financial toxicity in the past week. Will be assessed using mixed-effect analysis of variance to model the correlations.
Quality of life (QOL) | At T0 (3 months) and T1 (3 months post-intervention)
  Will be measured by the European QoL 5-Dimension questionnaire (EQ-5D), a widely used instrument to measure patients' QOL. The EQ-5D is a 2-part questionnaire. Will be calculated based on the technique of composite time trade-off preferences and scores of the 5 domains, indicating that -0.573 = worst health and 1 = best health. Will be assessed using mixed-effect analysis of variance to model the correlations.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbing Bai, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (4):
- United States (4):
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia